CLINICAL TRIAL: NCT06529042
Title: Prediction of Adverse Outcomes in Pregnancies of Individuals With Sickle Cell Disease - SCRIPT: Sickle Cell Risk in Pregnancy Tool
Brief Title: SCRIPT: Sickle Cell Risk in Pregnancy Tool
Acronym: SCRIPT
Status: Enrolling by invitation | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Johns Hopkins University (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); St. Paul's Hospital, Vancouver (Providence Health Care) (Unknown)
Responsible Party: Sponsor
Other Study IDs: SCRIPT
Record Dates: First submitted 2024-06-26; First posted 2024-07-31 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease; Pregnancy, High Risk; Pregnancy Complications
Keywords: Risk Assessment; Bayesian Prediction
MeSH Terms: conditions — Anemia, Sickle Cell; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnancies of Individuals with Sickle Cell Disease
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
Sickle Cell Disease (SCD), common in persons of Black ancestry, affects the shape of hemoglobin, the oxygen-carrying part of red blood cells (RBC). It is characterized by many complications, the most dreaded of which are related to pregnancy - affecting both the mother and unborn child. Compared to those without SCD, people with SCD have more adverse pregnancy outcomes (APO): 6x maternal mortality, 2x preeclampsia & preterm birth, 4x risk of having a baby not growing well in the womb & stillbirth. There is also greater need for access to care (7x higher hospitalization often multiple times lasting days to months). Yet up to 30% of SCD pregnancies are uncomplicated.

Treatments in pregnancy are limited and carry risks. A method to distinguish pregnancies at high-risk of APO that may benefit from these potentially risky treatments, from those likely to be uncomplicated, is urgently needed. To meet this need, the investigators developed a calculator to estimate pregnancy complication risk, using single-centre data. Its accuracy and precision will now be evaluated with international information from several centers by testing the calculator, and adjusting it as needed, using already available pregnancy-data from study centres in several countries. Those age >16 years, who have a confirmed SCD genotype, pregnancy with one baby, and pregnancy care and birth at a participating study centre will be included. Pregnancy care for the participants will be up to their doctors, with no changes based on the study. SCRIPT - the new tool - will guide future care by predicting who may benefit from specific treatments, reducing harm to low-risk individuals & will allow selection of high-risk patients for a future trials to determine whether currently available and novel treatments in well-selected patients can improve APO sufficiently to balance treatment-related harms.

DETAILED DESCRIPTION:
Sickle Cell Disease (SCD) is the most common haemoglobinopathy; predominantly affecting persons of African descent(1). In comparison to those without SCD, pregnant persons with SCD have a six-fold higher risk of mortality, twice the risk of preeclampsia and preterm birth, and nearly a four-fold risk of having a small for gestational age infant or experiencing stillbirth(2,3). Furthermore, there is a higher rate of resource utilization in this group, with nearly 50% of pregnancies complicated by at least one antenatal admission and an overall seven-fold higher hospitalization risk compared to pregnancies without SCD(4,5). These admissions are most commonly secondary to vaso-occlusive events or anemia, can occur on multiple occasions, and can last days to months(4,5).

During pregnancy, red blood cell (RBC) transfusion remains the only recommended intervention(6), with some evidence suggesting that prophylactic transfusion may modify adverse pregnancy outcomes (APOs)(7,8), with a possible positive effect on hospitalization rates through decreased complications, though this requires further study. However, transfusion is not without risk. Beyond its typically-feared infectious complications(9), transfusion in SCD is associated with alloimmunization rates of over 30%(10-12), can induce life-threatening hyperhemolysis(13), and will eventually lead to iron overload(14). At the same time, up to 30% of pregnancies in individuals with SCD remain uncomplicated(2,3,15,16).

A tool is thus urgently needed to separate high-risk individuals who would benefit from transfusion from low-risk individuals who would accrue transfusion risks with minimal, if any benefit. Using a single-centre cohort, the investigators developed maternal and fetal risk prediction models, as the first step in permitting the selection of patients most likely to benefit from transfusion(16). Ultimately, a multi-center international randomized controlled trial (RCT) is required to determine the benefits of prophylactic transfusion in this setting; yet, before such an RCT is conceived, the model(s) must be refined and validated with a larger sample to allow for appropriate participant selection.

The investigators proposed a multicenter international cohort study to enhance the predictive capacity and validate the current model(s) within the participating centers. The academic centers (located in Canada, USA, and France), have multi-disciplinary experts dedicated to managing pregnant persons with SCD, and the combination of MFM and Haematology site co-leads provides essential interdisciplinary expertise with synergistic medical and obstetric perspectives.

Once completed, the Sickle Cell Risk In Pregnancy Tool (SCRIPT) will inform medical decisions regarding transfusion and will set the stage for appropriate selection of high-risk individuals for inclusion in an RCT aimed to definitively determine whether prophylactic transfusion in well-selected pregnant individuals with SCD does indeed improve APOs to the degree that would balance its potential associated harms.

ELIGIBILITY:
Inclusion Criteria:

* Age >16 years
* HbSS, HbSC, HbS/β0-thalassemia, HbS/β+-thalassemia confirmed on Hb electrophoresis, high performance liquid chromatography, capillary electrophoresis, or genetic testing
* Records of pregnancy care and birth at a participating centre
* Pregnancy continuing to at least 16+0 weeks' gestation (41,42)

Exclusion Criteria:

* Inability to confirm SCD genotype
* Incomplete medical records.

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant Individuals with Sickle Cell Disease (HbSS, HbSC, HbS/β0-thalassemia, HbS/β+-thalassemia)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of Adverse Pregnancy Outcome | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of the following events first noted during the pregnancy within the study period: acute anemia (yes, no), cardiac complication (yes, no), pulmonary complication (yes, no), hepatobiliary complication (yes, no), MSK complication (yes, no), splenic complication (yes, no), neurologic complication (yes, no), renal complication (yes, no); multi-organ failure (yes, no), venous thromboembolism (yes, no), vaso-occlusive event with admission (yes, no), red cell transfusion (yes, no), maternal mortality (yes, no), hypertensive disorder of pregnancy (yes, no), preterm birth (yes, no), small for gestational age (yes, no), or perinatal mortality (yes, no); defined based on published classifications.

SECONDARY OUTCOMES:
Presence of Acute Anemia | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: hyperhemolysis [clinical diagnosis], acute splenic sequestration; hepatic sequestration, or aplastic crisis; defined based on published classification
Presence of Cardiac Complications | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: congestive heart failure, cardiomyopathy, cardiomegaly, or arrhythmia; defined based on published classification
Presence of Pulmonary Complications | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: acute chest syndrome; pneumonia, or pulmonary hypertension; defined based on published classification
Presence of Hepato-Biliary Complications | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: cholecystitis, cholelithiasis; cholecystectomy; cholestasis of pregnancy, or viral hepatitis; defined based on published classification
Presence of Musculo-Skeletal Complications | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: avascular necrosis, ulcer, myositis, or osteomyelitis; defined based on published classification
Presence of Neurologic Complications | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: silent cerebral infarct, cerebrovascular accident, cerebral aneurysm, transient ischemic attack, or Moya-Moya syndrome; defined based on published classification
Presence of Renal Complications | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: acute kidney injury, proteinuria, pyelonephritis, or hematuria; defined based on published classification
Presence of Multi-Organ Failure | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Consultant's opinion in chart note specifying a diagnosis of "MOF" during current study pregnancy; clinical diagnosis
Presence of Venous Thromboembolism | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: deep vein thrombosis, pulmonary embolism, atypical site venous thrombosis, or cerebral venous sinus thrombosis (CVST); defined based on published classification
Presence of Vaso-Occlusive Event with Admission | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Vaso-Occlusive Event (VOE): New onset pain lasting >4 hrs in current study pregnancy, for which there is no explanation other than vaso-occlusion, and which requires presentation for acute care - patient self-report
Provision of Red Blood Cell Transfusion | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: simple transfusion in pregnancy, exchange transfusion (manual exchange or erythrocytapheresis), or prophylactic transfusion
Occurrence of Maternal Mortality | During pregnancy (until delivery of infant, up to 42 weeks of gestation) and continuing to 6 months postpartum
  Maternal death during current study pregnancy and up to 6 months postpartum
Presence of Hypertensive Disorder of Pregnancy | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Yes, if any of: Gestational Hypertension (gHTN) [persistent de novo HTN over 20 weeks' GA in absence of features of preeclampsia], Pre-eclampsia (PET) [gHTN + >1 new onset conditions >20 weeks GA - proteinuria or maternal organ/uteroplacental dysfunction], Eclampsia [new onset seizures in context of pre-eclampsia]; or HELLP Syndrome [Evidence of Hemolysis, Elevated Liver Enzymes, Low Platelets in context of pre-eclampsia]
Occurrence of Preterm Birth | During pregnancy (until delivery of infant, up to 42 weeks of gestation)
  Preterm birth (< 37+0 weeks GA) during current study pregnancy
Presence of Small for Gestational Age (SGA) Size | At delivery of infant
  Birthweight <10th centile for gestational age
Occurrence of Perinatal Mortality | During pregnancy (until delivery of infant, up to 42 weeks of gestation) and up to 28 days after birth)
  Intrauterine fetal demise (IUFD) [absence of FHR at or after 20 weeks' gestation] or Neonatal Death (NND) [death before 28 days of life, following live birth]

CONTACTS AND LOCATIONS:
Overall Officials: A. Kinga Malinowski, MD, MSc, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (3):
- Johns Hopkins University, Baltimore, Maryland, United States
- Canada (2):
  - Providence Health Care, Vancouver, British Columbia
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boafor TK, Olayemi E, Galadanci N, Hayfron-Benjamin C, Dei-Adomakoh Y, Segbefia C, Kassim AA, Aliyu MH, Galadanci H, Tuuli MG, Rodeghier M, DeBaun MR, Oppong SA. Pregnancy outcomes in women with sickle-cell disease in low and high income countries: a systematic review and meta-analysis. BJOG. 2016 Apr;123(5):691-8. doi: 10.1111/1471-0528.13786. Epub 2015 Dec 15. PMID 26667608
- [Background] Oteng-Ntim E, Meeks D, Seed PT, Webster L, Howard J, Doyle P, Chappell LC. Adverse maternal and perinatal outcomes in pregnant women with sickle cell disease: systematic review and meta-analysis. Blood. 2015 May 21;125(21):3316-25. doi: 10.1182/blood-2014-11-607317. Epub 2015 Mar 23. PMID 25800049
- [Background] Sun PM, Wilburn W, Raynor BD, Jamieson D. Sickle cell disease in pregnancy: twenty years of experience at Grady Memorial Hospital, Atlanta, Georgia. Am J Obstet Gynecol. 2001 May;184(6):1127-30. doi: 10.1067/mob.2001.115477. PMID 11349177
- [Background] Yu CK, Stasiowska E, Stephens A, Awogbade M, Davies A. Outcome of pregnancy in sickle cell disease patients attending a combined obstetric and haematology clinic. J Obstet Gynaecol. 2009 Aug;29(6):512-6. doi: 10.1080/01443610903003175. PMID 19697199
- [Background] Chou ST, Alsawas M, Fasano RM, Field JJ, Hendrickson JE, Howard J, Kameka M, Kwiatkowski JL, Pirenne F, Shi PA, Stowell SR, Thein SL, Westhoff CM, Wong TE, Akl EA. American Society of Hematology 2020 guidelines for sickle cell disease: transfusion support. Blood Adv. 2020 Jan 28;4(2):327-355. doi: 10.1182/bloodadvances.2019001143. PMID 31985807
- [Background] Malinowski AK, Shehata N, D'Souza R, Kuo KH, Ward R, Shah PS, Murphy K. Prophylactic transfusion for pregnant women with sickle cell disease: a systematic review and meta-analysis. Blood. 2015 Nov 19;126(21):2424-35; quiz 2437. doi: 10.1182/blood-2015-06-649319. Epub 2015 Aug 24. PMID 26302758
- [Background] Vianello A, Vencato E, Cantini M, Zanconato G, Manfrin E, Zamo A, Zorzi F, Mazzi F, Martinelli N, Cavaliere E, Monari F, Venturelli D, Ferrara F, Olivieri O, De Franceschi L. Improvement of maternal and fetal outcomes in women with sickle cell disease treated with early prophylactic erythrocytapheresis. Transfusion. 2018 Sep;58(9):2192-2201. doi: 10.1111/trf.14767. Epub 2018 Jul 8. PMID 29984534
- [Background] Chou ST. Transfusion therapy for sickle cell disease: a balancing act. Hematology Am Soc Hematol Educ Program. 2013;2013:439-46. doi: 10.1182/asheducation-2013.1.439. PMID 24319217
- [Background] Kacker S, Ness PM, Savage WJ, Frick KD, Shirey RS, King KE, Tobian AA. Economic evaluation of a hypothetical screening assay for alloimmunization risk among transfused patients with sickle cell disease. Transfusion. 2014 Aug;54(8):2034-44. doi: 10.1111/trf.12585. Epub 2014 Feb 27. PMID 24571485
- [Background] Yazdanbakhsh K, Ware RE, Noizat-Pirenne F. Red blood cell alloimmunization in sickle cell disease: pathophysiology, risk factors, and transfusion management. Blood. 2012 Jul 19;120(3):528-37. doi: 10.1182/blood-2011-11-327361. Epub 2012 May 4. PMID 22563085
- [Background] Balbuena-Merle R, Hendrickson JE. Red blood cell alloimmunization and delayed hemolytic transfusion reactions in patients with sickle cell disease. Transfus Clin Biol. 2019 May;26(2):112-115. doi: 10.1016/j.tracli.2019.02.003. Epub 2019 Feb 22. PMID 30857806
- [Background] Danaee A, Inusa B, Howard J, Robinson S. Hyperhemolysis in Patients With Hemoglobinopathies: A Single-Center Experience and Review of the Literature. Transfus Med Rev. 2015 Oct;29(4):220-30. doi: 10.1016/j.tmrv.2015.06.001. Epub 2015 Jun 19. PMID 26209603
- [Background] Tavares AHJ, Benites BD, Fertrin KY. Myocardial Iron Overload in Sickle Cell Disease: A Rare But Potentially Fatal Complication of Transfusion. Transfus Med Rev. 2019 Jul;33(3):170-175. doi: 10.1016/j.tmrv.2019.04.001. Epub 2019 May 2. PMID 31153715
- [Background] Silva FAC, Ferreira ALCG, Hazin-Costa MF, Dias MLG, Araujo AS, Souza AI. Adverse clinical and obstetric outcomes among pregnant women with different sickle cell disease genotypes. Int J Gynaecol Obstet. 2018 Oct;143(1):89-93. doi: 10.1002/ijgo.12626. Epub 2018 Aug 6. PMID 30030929
- [Background] Malinowski AK, Kuo KHM, Tomlinson GA, Palcu P, Ward R, Shehata N. Distinct maternal and fetal pregnancy outcomes in women with sickle cell disease can be predicted using routine clinical and laboratory data. Br J Haematol. 2021 Sep;194(6):1063-1073. doi: 10.1111/bjh.17607. Epub 2021 Jun 14. PMID 34124774
- [Background] Odendaal H, Wright C, Brink L, Schubert P, Geldenhuys E, Groenewald C. Association of late second trimester miscarriages with placental histology and autopsy findings. Eur J Obstet Gynecol Reprod Biol. 2019 Dec;243:32-35. doi: 10.1016/j.ejogrb.2019.10.024. Epub 2019 Oct 22. PMID 31670146
- [Background] Roberge S, Nicolaides KH, Demers S, Villa P, Bujold E. Prevention of perinatal death and adverse perinatal outcome using low-dose aspirin: a meta-analysis. Ultrasound Obstet Gynecol. 2013 May;41(5):491-9. doi: 10.1002/uog.12421. PMID 23362106
- [Background] Ballas SK, Lieff S, Benjamin LJ, Dampier CD, Heeney MM, Hoppe C, Johnson CS, Rogers ZR, Smith-Whitley K, Wang WC, Telen MJ; Investigators, Comprehensive Sickle Cell Centers. Definitions of the phenotypic manifestations of sickle cell disease. Am J Hematol. 2010 Jan;85(1):6-13. doi: 10.1002/ajh.21550. PMID 19902523
- [Background] Magee LA, Pels A, Helewa M, Rey E, von Dadelszen P; Canadian Hypertensive Disorders of Pregnancy Working Group. Diagnosis, evaluation, and management of the hypertensive disorders of pregnancy: executive summary. J Obstet Gynaecol Can. 2014 May;36(5):416-41. doi: 10.1016/s1701-2163(15)30588-0. English, French. PMID 24927294
- [Background] Kramer MS, Platt RW, Wen SW, Joseph KS, Allen A, Abrahamowicz M, Blondel B, Breart G; Fetal/Infant Health Study Group of the Canadian Perinatal Surveillance System. A new and improved population-based Canadian reference for birth weight for gestational age. Pediatrics. 2001 Aug;108(2):E35. doi: 10.1542/peds.108.2.e35. PMID 11483845